CLINICAL TRIAL: NCT06127927
Title: Evaluation the Efficacy and Safety of an Interventional Left Ventricular Assist System for Hemodynamic Support in Patients With Cardiogenic Shock: A Prospective, Multicenter, Single-group Target Value Study of Sustained
Brief Title: An Interventional Left Ventricular Assist System for Cardiogenic Shock
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Liang-Wan Chen MD, Chief, Fujian Medical University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A202301
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Cardiogenic Shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Left Ventricular Assist System Pre-trial (Experimental): The design of the first phase pre-trial clinical study will involve a total of 6 subjects. The survival rate of subjects before discharge or 30 days after weaning was the main effectiveness evaluation indicator, and the safety and effectiveness of the test device were preliminarily evaluated. All SAE events during the study will be reviewed by CEC experts. According to the expert review opinions, if no unexpected serious complications and product defects are found, the Formal Research phase will be started.
  Interventions: Device: Interventional Left Ventricular Assist System
- Interventional Left Ventricular Assist System Formal Research (Experimental): A formal clinical trial to evaluate the effectiveness and safety of interventional left ventricular assist system for hemodynamic support in patients with cardiogenic shock through a prospective, multicenter, single-group target value study.The total number of patients enrolled in this study is planned to be 54. This sample size is calculated according to statistical principles, combining the research hypothesis and the estimate of the expected level of efficacy. The sample size calculation is based on the main efficacy index and the main safety index. Since it is set according to the common evaluation index, the sample size is calculated for the two main evaluation indicators separately, and the largest one is used as the final sample size of this trial.
  Interventions: Device: Interventional Left Ventricular Assist System

INTERVENTIONS:
Device: Interventional Left Ventricular Assist System — Interventional left ventricular assist system for cardiogenic shock patients

SUMMARY:
Imported Impella The price is relatively expensive and difficult for ordinary patients to afford. In order to better meet the growing clinical needs in China, Anhui Tongling Bionic Technology Co., Ltd. has developed an interventional left ventricular assist system. The test device was tested in preclinical animals It has shown good effectiveness and safety. Through the implementation of this clinical trial, the interventional left ventricular assist system The safety and effectiveness of the system for hemodynamic support in patients with cardiogenic shock have led to further development of this product in the country.

DETAILED DESCRIPTION:
In recent years, patients with severe heart disease, with coronary heart disease as the main disease spectrum, have been on the rise, and the mortality rate remains high. In routine clinical diagnosis and treatment, inotropic drugs and vasoactive drugs are used to correct shock and maintain blood flow. The cornerstone of mechanical stability, however, there is insufficient evidence that these drugs benefit patients in the long term. Mechanical circulatory support (MCS) is a life support technology that was firstly used clinically in the 1950s. It can replace or partially replace the functions of the heart and/or lungs. And by increasing end-organ and coronary artery perfusion, reducing cardiac volume load, ventricular wall stress and myocardial oxygen consumption, etc. mechanism, quickly and accurately produce a stable hemodynamic effect, ultimately reducing the patient's pulmonary circulation congestion and myocardial ischemia. Reduce blood flow and infarction area and gain valuable time for follow-up treatment, so that patients with severe heart disease can be supported and transitioned to treatment great progress has been made in the treatment of heart diseases, and this technology has been widely used in the field of critical heart disease. 2017 American Heart Association The American Heart Association (AHA) recommends MCS for waiting for recovery of cardiac function or heart transplantation. Interimplantation and definitive treatment of advanced heart failure. Depending on location, MCS is divided into left ventricle Left ventricular assist device (LVAD), right ventricular assist device (Right ventricular assist device (RVAD), biventricular assist device (Biventricular assist device, BVAD) and total artificial heart (TAH). Currently, MCS commonly used in clinical practice mainly includes Intra-aortic balloon pump (IABP), extracorporeal membrane oxygenation (Extracorporeal membrane oxygenation (ECMO), Impella, TandemHeart and RVAD. The Impella system is an LVAD, it is divided into 3 models according to the diameter of the instrument: 12F (Impella 2.5), 14F (Impella CP) and 21F (Impella 5.0), the corresponding maximum output flows are 2.5L/min, 3.0~4.0L/min and 5.0L/min. The working principle of the device is to pump the left heart through the built-in micro axial flow pump at the front end of the catheter.

The oxygenated blood in the ventricle is pumped out through the catheter inlet, and then the axial flow pump is pumped directly into the ascending aorta to establish the left ventricular-ascending aorta. Aortic drainage pathway. Can help increase cardiac output (CO), increase aortic pressure and Coronary perfusion pressure, improve mean arterial pressure, coronary blood flow; while reducing left ventricular preload and pulmonary Pulse wedge pressure reduces ventricular wall tension and myocardial oxygen consumption. Acts as an active mechanical pump and partially replaces left ventricular function able. Impella is commonly used in the clinical treatment of cardiogenic shock. The ISAR-SHOCK study enrolled 26 patients with acute cardiac arrest. Comparing the efficacy of IABP and Impella 2.5 in patients with cardiogenic shock after myocardial infarction, the primary endpoint of the study Changes in cardiac index (CI) 30 minutes after MCS insertion. It was found that Impella A more significant increase in CI than after IABP, with 30-day mortality of 46% in both groups, confirms that Impella 2.5 Safety and feasibility in the treatment of cardiogenic shock after acute myocardial infarction. Two other studies also found that Similar conclusion RECOVER I study is a study that included 16 cases of cardiogenic shock or hypocardia after cardiotomy. A prospective, single-arm study of patients with displacement syndrome, the results of which indicate immediate blood loss after implantation of Impella 5.0 Fluid dynamics indicators improved significantly, and 93% of patients had improved cardiac function at discharge, with all patients at 30 days, 3 months, and 1 year. The survival rates were 94%, 81% and 75% respectively, proving the safety of Impella 5.0 for bridging treatment after cardiac surgery and feasibility. Currently, only Impella produced by the American company Abiomed has been approved by the FDA. However, imported Impella The price is relatively expensive and difficult for ordinary patients to afford. In order to better meet the growing clinical needs in China, Anhui Tongling Bionic Technology Co., Ltd. has developed an interventional left ventricular assist system. The test device was tested in preclinical animals It has shown good effectiveness and safety. Through the implementation of this clinical trial, the interventional left ventricular assist system The safety and effectiveness of the system for hemodynamic support in patients with cardiogenic shock have led to further development of this product in the country.

ELIGIBILITY:
For Pre-trial Phase

Inclusion Criteria:

1. Age 18-75 years old;
2. Refractory cardiogenic shock as determined by the cardiac MDT expert group; The criteria for refractory cardiogenic shock are: despite adequate doses of two vasoactive drugs and treatment of the underlying cause, there is still evidence of tissue hypoperfusion;
3. The subject can understand the purpose of the trial, voluntarily participate and sign the written informed consent form reviewed and approved by the ethics committee; the subject agrees to complete the follow-up in accordance with the protocol requirements.

Exclusion Criteria:

1. Right heart failure that meets any of the following conditions:

   a Central venous pressure-capillary wedge pressure ≥10mmHg; b Central venous pressure-pulmonary artery diastolic pressure ≥10mmHg; c Cardiac tamponade.
2. Any peripheral vascular disease that prevents the placement of the trial device;
3. Left or right ventricular thrombus;
4. Aortic valve regurgitation, echocardiographic grade ≥2+;
5. Aortic valve stenosis, valve area ≤1.5cm2;
6. Aortic valve calcification;
7. Presence of mechanical aortic valve;
8. Hypertrophic or obstructive cardiomyopathy;
9. Untreated ventricular septal or atrial septal defect;
10. Patent foramen ovale;
11. Mechanical complications of acute myocardial infarction;
12. Presence of hereditary spherocytosis, hereditary elliptocytosis, autoimmune hemolytic anemia or other diseases that cause hemolysis;
13. Cardiopulmonary resuscitation lasting more than 15 minutes within 24 hours before catheter pump implantation;
14. Ventricular tachycardia or ventricular fibrillation is ineffective with drug treatment;
15. Renal failure, serum creatinine ≥309.4umol/l or blood urea nitrogen ★ ≥35.7mmol/l);
16. Liver failure (total bilirubin ≥85.5umol/l);
17. Allergy or intolerance to heparin;
18. Presence of any cardiac assist device;
19. Presence of active systemic infection;
20. Refusing to sign the informed consent form or failing to complete follow-up as required by the protocol;
21. Pregnant or lactating women, female subjects with potential fertility but unable or unwilling to use effective contraceptive measures during the study;
22. Subjects who have participated in other clinical trials within 3 months or are currently participating in other clinical trials;
23. Other situations that the investigator believes are not suitable for clinical trials.

For Formal Research Phase

Inclusion Criteria:

1. Age 18-75 years old;
2. Low cardiac output syndrome or increased filling pressure after regular continuous pumping of 1 high-dose or 2 medium-dose inotropic drugs within 48 hours after cardiopulmonary bypass was removed during cardiac surgery. The specific criteria are as follows;

The drugs, doses and time of 1 high-dose or 2 medium-dose inotropic drugs are as follows:

Epinephrine: medium dose (<0.03 μg/kg/min), continuous pumping ≥15 minutes High dose (≥0.03 μg/kg/min), continuous pumping ≥15 minutes; Dobutamine: medium dose (<5μg/kg/min), continuous pumping ≥15 minutes High dose (≥5μg/kg/min), continuous pumping ≥15 minutes; Milrinone: medium dose (<0.3 μg/kg/min), continuous pumping ≥120 minutes High dose (≥0.3 μg/kg/min), continuous pumping ≥120 minutes; Low cardiac output syndrome: cardiac index 1.3≤CI≤2.2 L/min/m2;

Increased filling pressure: pulmonary capillary wedge pressure:

20≤PCWP≤30mmHg or pulmonary artery systolic pressure: 25≤PAP≤35mmHg 3) The subject can understand the purpose of the trial, voluntarily participate and sign the informed consent form reviewed and approved by the ethics committee; the subject agrees to complete the follow-up in accordance with the protocol requirements.

Exclusion Criteria:

1. Right heart failure that meets any of the following conditions:

   1. Central venous pressure-capillary wedge pressure ≥10mmHg;
   2. Central venous pressure-pulmonary artery diastolic pressure ≥10mmHg;
   3. Cardiac ascites.
2. Any peripheral vascular disease that prevents the placement of the trial device;
3. Left or right ventricular thrombus;
4. Aortic valve regurgitation, echocardiographic grade ≥2+;
5. Aortic valve stenosis, valve area ≤1.5cm2;
6. Presence of mechanical aortic valve;
7. Hypertrophic or obstructive cardiomyopathy;
8. Untreated ventricular septal or atrial septal defect;
9. Patent foramen ovale;
10. Mechanical complications of acute myocardial infarction;
11. Suffering from diseases that cause increased blood cell fragility or hemolysis;
12. Cardiopulmonary resuscitation lasting more than 15 minutes within 24 hours before catheter pump implantation;
13. Sustained or non-sustained ventricular tachycardia or ventricular fibrillation that is unresponsive to drug treatment;
14. Renal failure, serum creatinine ≥3.5mg/dl or blood urea nitrogen ≥100mg/dl;
15. Liver failure, total bilirubin ≥5mg/dl;
16. Allergy or intolerance to heparin;
17. Other cardiac assist devices other than IABP have been implanted;
18. Active systemic infection;
19. Refuse to sign the informed consent form or fail to complete follow-up as required by the protocol;
20. Pregnant or lactating women, female subjects with potential fertility but unable or unwilling to use effective contraceptive measures during the study;
21. Subjects who are participating in other clinical trials and have not yet reached the endpoints of the trial;
22. Other situations that the investigator believes are not suitable for clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-11-08 (Estimated); Study Completion 2025-12-08 (Estimated)

PRIMARY OUTCOMES:
Survival rate of subjects at discharge or 30 days after weaning from ventilator (whichever is longer) | 30days
  Survival was defined as recovery of cardiac function or survival to bridging therapy; Recovery of cardiac function was defined as no need for any mechanical support or IABP assistance 30 days after removal of the invasive left ventricular assist system or at discharge (whichever was longer).
  Survival to bridging therapy was defined as survival to the induction of anesthesia for heart transplantation or placement of an implantable ventricular assist device.
The incidence of major adverse events at discharge or 30 days after weaning (whichever is longer) | 30days
  Major adverse events included death and stroke.

SECONDARY OUTCOMES:
hemodynamic indicators | 30days
  Immediately after surgery, before weaning, and 24 hours after weaning, researchers evaluated the improvement in the subjects' hemodynamics after implantation of the trial device. (cardiac index(L/min/m2), mean arterial pressure(mmHg), pulmonary diastolic pressure(mmHg))
Successful device placement and technical success | 30days
  Successful device placement is defined as the successful placement of a disposable left ventricular catheter pump into the left ventricle via the artery, and the delivery system can be withdrawn smoothly.
  Technical success: After successful placement of the test device, blood can be pumped from the left ventricle into the ascending aorta, increasing the subject's cardiac output.

CONTACTS AND LOCATIONS:
Overall Officials: Liang-wan Chen, M.D Ph.D, Study Chair — Fujian Medical University Union Hospital
Locations (2):
- China (2):
  - Department of Cardiovascular Surgery, Fuzhou, Fujian
  - Fujian Medical University Union Hospital, Fuzhou, Fujian

IPD SHARING:
Plan to Share IPD: No